CLINICAL TRIAL: NCT04973215
Title: HealthIntro - a Study to Increase the Successful Participation of Refugees With Health Problems in the Introduction Program
Brief Title: HealthIntro - Health Perspective in the Introduction Program
Acronym: HealthIntro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Tromso (Other)
Collaborators: NORCE Norwegian Research Centre AS (Other); FAFO Research foundation (Unknown); Harstad municipality (Unknown); Senja municipality (Unknown); Sør-Varanger municipality (Unknown)
Responsible Party: Principal Investigator, Johanna Laue, associate professor, University of Tromso
Other Study IDs: 237875
Record Dates: First submitted 2021-06-23; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Refugee Health
Keywords: immigration; refugees; introduction program; health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- work package 1: all participants in Norwegian introduction program and their family relations
  Interventions: Other: no intervention
- work package 2: strategic sample of refugees with health problems currently participating in the introduction program
  Interventions: Other: no intervention
- work package 3: 3-6 families from which one or more participate in the introduction program and one or more have health problems
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is not an intervention study

SUMMARY:
Health problems seem one major reason for why not all refugees, especially women, fulfill the introduction program (IP) and enter the labour market after the end of the program. This challenges integration, and can lead to increased inequalities in society. The HealthIntro pilot-project and existing knowledge point towards a mismatch between the IP's goal to integrate as many refugees as possible into the labour market as soon as possible, and the demanding situation refugees with complex (health) challenges face after resettlement in the host country. Particular barriers seem related to the little flexibility of the introduction law, difficulties with collaboration between public services and with involving refugees in decision-making regarding program adjustments. It is known that refugees have more health problems than the rest of the population. Additionally, current trends in integration policy result in increasing numbers of refugees with complex challenges in municipalities, often families in which one or several members have health problems. It is therefore of high importance to develop strategies that enable municipalities to work more effectively with these most vulnerable group of refugees in the early phase of resettlement and during the IP.

In collaboration with three North Norwegian municipalities and refugees, the investigators will explore how health problems interconnect with program participation on the national level, the municipal level and in a family context. Moreover, the investigators will use this knowledge to collaboratively generate ideas on how to improve the strategic work in municipalities with refugees with health problems. More specifically, the investigators will link registerdata on a national level, conduct explorative qualitative studies addressing the system level in municipalities, and the family and everday life context of refugee families, and conduct an action research inspired study to initiating change in municipalities.

DETAILED DESCRIPTION:
This study is funded by The Norwegian Research Council (project number 319050)

ELIGIBILITY:
Work package 1:

Inclusion criteria:

* refugee status
* participate or have participated in the introduction program in Norway

Exclusion criteria

* not refugee status
* not participated in the introduction program in Norway

Work package 2:

Inclusion criteria, sample 1

* refugee status
* participate in the introduction program in Harstad, Senja, or Sør-Varanger municipality during the project period and since at least one year at enrollment
* have a self-reported health problem

Exclusion criteria, sample 1

* no refugee status
* do not participate in the introduction program
* do not have a health problem

Inclusion criteria, sample 2

* has professional experience with refugees in Harstad, Senja, or Sør-Varanger municipality
* currently working in Harstad, Senja, or Sør-Varanger municipality
* above 18 years of age

Exclusion criteria, sample 2

* under 18 years of age
* not currently working in Harstad, Senja, or Sør-Varanger municipality

Work package 3:

Inclusion criteria:

* refugee status
* living together with family including one or more children
* participate in the introduction program in Harstad, Senja, or Sør-Varanger municipality during the project period and since at least one year at enrollment
* have a self-reported health problem within the family

Exclusion criteria_

* no refugee status
* do not participate in the introduction program
* do not live together with family
* do not have a health problem within the family

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Work package 1: all participants in the introduction program, since start of the program in Norway, and their family relations.
  Work package 2: persons with refugee status settled in Harstad, Senja, or Sør-Varanger municipality who participate in the introduction program during the project period and have a self-reported health problem (sample 1), employees working in Harstad, Senja, or Sør-Varanger municipality with experience with refugees and the introduction program during their work
  Work package 3: families with refugee status settled in Harstad, Senja, or Sør-Varanger municipality, which have one or several health problems within the family and of which one or both parents participate in the introduction program.
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Work package 1: Number of refugees dropping out of the introduction program or being unemployed after the end of the program; diagnoses associated with drop out of the program . | WP 1: 5-10 years after having finished the introduction program
  Work packages 2-4 are qualitative studies and cannot be described in terms of outcome measures due to methodological reasons

IPD SHARING:
Plan to Share IPD: No